CLINICAL TRIAL: NCT01198847
Title: A Randomised Controlled Trial for Overweight and Obese Parents to Prevent Childhood Obesity
Brief Title: Early Stockholm Obesity Prevention Program
Acronym: EarlySTOPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Claude Marcus, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ES-2010
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Obesity; Overweight
Keywords: child overweight; child obesity; prevention; targeted intervention; development of overweight
MeSH Terms: conditions — Obesity; Overweight; Pediatric Obesity | interventions — Diet; Exercise; Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low intensity arm (Active Comparator): Written information about a healthy lifestyle
  Interventions: Behavioral: Dietary, physical activity and sleeping
- High intensity arm (Experimental): Lifestyle support (PA, sleep, food intake) using MI
  Interventions: Behavioral: Dietary, physical activity and sleeping

INTERVENTIONS:
Behavioral: Dietary, physical activity and sleeping — The intervention in the present study will be delivered through sessions aiming at developing healthy lifestyle habits regarding physical activity, food intake and regular sleeping habits for parents and children. These sessions will be performed face to face by trained health care workers and carried out in the welfare centres with the parent/s. Children will not be approached directly in the present study. All families will meet with their coach/facilitator during at least 12 times (including start and final evaluation meeting) until the children reach 6 years of age (such as school age). However extra effort (as boosting sessions) will be made if growth records show an increased BMI (weight induced meetings). The parents are also encouraged to keep contact with their coach either by phone or e-mail as often as they feel needed.
  The Low intensity arm will only receive written information and no direct face to face support

SUMMARY:
To study whether a targeted intervention can prevent the development of overweight and obesity among pre-school children in families with either one obese or two overweight parents.

DETAILED DESCRIPTION:
Early STOPP project wants to promote good health in children from early age by supporting good habits for the whole family. Our aim is to see if we can prevent overweight and obesity in children in families where parents are overweight or obese. Normal weight parents will also be needed in this study.

Background Life is in constant change and affects our habits. In many ways this is positive but it also contributes to less favorable health factors. For example, take the car instead of cycling, take the lift instead of the stairs. This makes us less active in everyday life. Individuals also eat more unhealthy foods in larger portions. In combination with genetics, social in heritage and surrounding factors this contributes to increase overweight and obesity among children not only in adults but also in children.

Good treatment methods for childhood obesity are lacking, making prevention very important. The earlier good habits are introduced to a child the better it is.

In Early STOPP project we study food, physical activity and sleep habits in the families with a little child. The height, weight, waist circumference and blood pressure will be recorded in both child and parents. The parents will answer questionnaires about food, physical activity and sleeping habits for both the child and themselves. During the study, the child's physical activity will be measured.

ELIGIBILITY:
Inclusion Criteria:

* one obese or two overweight parents, 1 year old child

Exclusion Criteria:

* weight effecting diseases

Ages: 1 Year to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 195 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Body Mass Index score(BMI sds) at the age 6 years to monitor the effectiveness of the intervention | 5 years
  Weight gain, reflected in BMI sds will reflect if the intervention has been successful

SECONDARY OUTCOMES:
sleeping behavior | 5 years
  sleeping duration will be monitored to study its effect on intervention
biomarkers | 5 years
  such as bacterial population in feces, markers in blood and in saliva
physical activity and sedentary behaviour | 5 years
  physical activity and sedentary behavious will be monitored during the intervention
dietary intake | 5 years
  changes in dietary habits and behaviour will be monitored
socioeconomic factors | 5 years
  factors effecting obesity development will be assessed in order to understand their impact on intervention

CONTACTS AND LOCATIONS:
Overall Officials: claude marcus, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Stcokholm, Sweden

REFERENCES:
- [Background] Sobko T, Svensson V, Ek A, Ekstedt M, Karlsson H, Johansson E, Cao Y, Hagstromer M, Marcus C. A randomised controlled trial for overweight and obese parents to prevent childhood obesity--Early STOPP (STockholm Obesity Prevention Program). BMC Public Health. 2011 May 18;11:336. doi: 10.1186/1471-2458-11-336. PMID 21592388
- [Derived] Bergqvist-Noren L, Hagman E, Xiu L, Marcus C, Hagstromer M. Physical activity in early childhood: a five-year longitudinal analysis of patterns and correlates. Int J Behav Nutr Phys Act. 2022 Apr 20;19(1):47. doi: 10.1186/s12966-022-01289-x. PMID 35443696
- [Derived] Xiu L, Ekstedt M, Hagstromer M, Bruni O, Bergqvist-Noren L, Marcus C. Sleep and Adiposity in Children From 2 to 6 Years of Age. Pediatrics. 2020 Mar;145(3):e20191420. doi: 10.1542/peds.2019-1420. Epub 2020 Feb 18. PMID 32071262
- [Derived] Johansson E, Hagstromer M, Svensson V, Ek A, Forssen M, Nero H, Marcus C. Objectively measured physical activity in two-year-old children - levels, patterns and correlates. Int J Behav Nutr Phys Act. 2015 Jan 24;12:3. doi: 10.1186/s12966-015-0161-0. PMID 25616495